Protocol ID: R44HD082968

ClinicalTrials.gov ID: NCT03655951
Title: Birds and Bees Research Study
Contact: Dr. Tracy Scull (tscull@irtinc.us)

IRB Reviewed Protocol - last updated approval date: 11/30/2018

## **Study Protocol and Statistical Analysis Plan**

The goal of this efficacy study was to evaluate how *Media Aware Parent*, a web-based program for parents to promote adolescent sexual health, influence parents' and children's sexual health knowledge; attitudes, efficacy, intentions, and behaviors about parent-adolescent communication; attitudes about media messages; and media message deconstruction skills. Parent consumer satisfaction with the program was also assessed. An Institutional Review Board approved of the methods and measures used in this study. The procedure used for conducting the research study is as follows:

- 1. Parents were recruited through a website and flyers that advertised this as a study where parents would be asked to evaluate online resources that could be helpful in talking about sexual health with their child. Inclusion criteria stipulated that participants be the parent or caregiver of a child in 7<sup>th</sup>, 8<sup>th</sup>, or 9<sup>th</sup> grade. Participants were also required to be proficient in English and have access to a laptop or tablet that had Wi-Fi capabilities (in order to access the study questionnaires and webbased resources). Those interested completed an online screener to determine their eligibility, and if eligible were then prompted to endorse online informed consent forms. Potential participants' information was verified by phone.
- 2. After a potential participant was recruited and verified, and if there was space in the study, the parent-child dyad was randomly assigned to condition 1) *Media Aware Parent* (intervention) or 2) active control. Group assignment was stratified by parent gender, race, and ethnicity.
- 3. Enrolled parents received two emails indicating that the family had been enrolled in the study, each including a link to access the pre-test questionnaires one for the parent and one for the child. Both had one week to complete their individual pretest questionnaires.
- 4. Parents received a reminder email, phone call, or text to complete the pretest questionnaires if both were not completed within 4 days of receiving access to the pretest questionnaire.
- 5. Parents also received a final reminder email, phone call, or text to complete the pretest questionnaires if both were not completed within 6 days of receiving access to the pretest questionnaire.

- 6. If both questionnaires were not completed after one week (7 days after enrollment), someone from the waitlist that could replace them (matched on gender, race, and ethnicity) was enrolled in the study.
- 7. Families that completed both of their pretest questionnaires received a \$30 Amazon.com gift card.
- 8. Upon completion of the pretest questionnaires, parents received a message at the end of the questionnaire informing them of their next steps in the research study. Parents in the intervention group learned that they will be asked to review Media Aware Parent. Parents in the control group learned that they will be asked to review online, CDC sexual health materials. Both groups were told they have two weeks (from the time both pretests have been completed) to review their materials to receive the program review incentive and that they will have the ability to revisit the resource during the duration of the study.
- 9. Parents were emailed with a link to their assigned resource.
- 10. All parents received a reminder after one week of receiving access to their resources to complete their review within the following week. All parents received a final reminder on about the 13<sup>th</sup> day to complete their review of the resource.
- 11. Four weeks after both pretest questionnaires were completed, parents received two emails with two links to access to the posttest questionnaires for both parent and child.
- 12. Parents received a reminder email, phone call, or text to complete the posttest questionnaires if both were not completed within 4 days of receiving access to the posttest.
- 13. Parents received a final reminder email, phone call, or text to complete the posttest questionnaires if both are not completed within 6 days of receiving access to the posttest.
- 14. Families that completed their resource review in the two-week timeframe and posttest questionnaires were emailed a \$95 Amazon.com gift card (\$45 for completing the resource review and \$50 for completing both second questionnaires).
- 15. Approximately 2-3 months after the posttest, we reached out to families via a mailed card to ask them to update their email address if it had changed.
- 16. About two to four weeks before a participant family was slated for the follow-up questionnaire, we sent a reminder of the upcoming final phase of the study.
- 17. Approximately six months after the pretest, parents received two emails with two links to access the follow-up questionnaires for the parent and child.
- 18. Parents received a reminder email to complete the follow-up questionnaires if both were not completed with 4 days of receiving access to the follow-up questionnaires.

- 19. Parents received a final reminder email to complete the follow-up questionnaires if both were not completed with 6 days of receiving access to the follow-up questionnaires.
- 20. Families that completed both their follow-up questionnaires were emailed a \$70 Amazon.com gift card.
- 21. Control parents were provided with access to Media Aware Parent after the study was completed.

## **Statistical Analyses Plan**

**Preliminary Analyses.** Psychometric analyses were conducted to confirm the reliability, validity, and distributions of key variables. To establish if there is baseline equivalence between groups, we tested for equivalence on basic demographic characteristics (i.e., age, race/ethnicity, gender, and sexual orientation) and on baseline levels of our primary outcome variables in a series of one-way ANOVA and  $\chi^2$  tests.

**Descriptive Statistics.** Interscale correlations were examined for the antecedent variables and outcome variables. Means, standard deviations, and ranges were calculated for the antecedent and outcome variables.

Main Analyses. To examine intervention effects, a residual difference score approach was used to provide an estimate of change from baseline (Little, 2013) and was assessed by regressing post-intervention scores onto baseline scores and the treatment variables. Binary outcomes were assessed with logistic regression. All analyses used standard errors which were robust to non-normality and heteroskedasticity and included gender, age, race, and ethnicity (for both parents and youth); youth's rating of parental relationship quality; and parent's religiosity as covariates. Missing data were handled using listwise deletion, also known as complete case analysis.